CLINICAL TRIAL: NCT04868864
Title: The Ontario Multi-Regional Hospital COVID-19 Registry (COREG)- Recovery Trajectory Sub-study
Acronym: COREG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, MyLinh Duong, Professor Department of Medicine, Hamilton Health Sciences Corporation
Organization: McMaster University (Other)
Other Study IDs: 13161
Record Dates: First submitted 2021-04-24; First posted 2021-05-03 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia; Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Tomography, X-Ray Computed; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate to severe COVID-19 infection: COVID-19 patients with radiographic changes on CXR or CT which had not resolved or had persistent hypoxia due to COVID-19 at the time of discharge will be enrolled. All participants will undergo a LDCT and PFT.
  Interventions: Diagnostic Test: CT scan; Diagnostic Test: Pulmonary Function Test
- Persistent LDCT or PFT abnormalities: Participants with abnormalities on LDCT and or PFT will be invited to continue with a follow-up sub-study. This will involve follow up with repeated LDCT and PFT at subsequent time points to monitor and manage the abnormalities detected until the abnormalities fully resolve or to the last time point at 9 months of the study.
  Interventions: Diagnostic Test: CT scan; Diagnostic Test: Pulmonary Function Test

INTERVENTIONS:
Diagnostic Test: CT scan — Non-enhanced LDCT scans of the thorax will be taken using standard technology on helical CT system
Diagnostic Test: Pulmonary Function Test — Standard pulmonary function testing will be conducted by trained pulmonary technologists following the American Thoracic Society standards

SUMMARY:
Radiological and lung function recovery following Covid-19 infection.

DETAILED DESCRIPTION:
The investigators propose to conduct pulmonary LDCT imaging and physiological lung function assessments, and combine this with detailed multi-regional hospitalization clinical data collection on COVID-19 cases (COREG registry); to inform long-term pulmonary and extra-pulmonary consequences and the recovery trajectory following COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from hospital post COVID-19 infection who have radiographic and clinical evidence of COVID-19 pneumonia during hospitalization.
* Patients with evidence of unresolved radiographic changes or persistent hypoxemia.

Exclusion Criteria:

* Failure to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients discharged from hospitals with radiographic and clinical evidence of COVID-19 pneumonia during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary changes on LDCT Scan | Through study completion, an average of 9 months
  Identify pulmonary changes utilizing LDCT chest to characterize the pulmonary recovery trajectory of survivors of COVID-19.

SECONDARY OUTCOMES:
DLCO | Through study completion, an average of 9 months
  Identify DLCO changes over time to characterize the pulmonary recovery trajectory of survivors of COVID-19.
TLC | Through study completion, an average of 9 months
  Identify TLC changes over time to characterize the pulmonary recovery trajectory of survivors of COVID-19.
FEV1 | Through study completion, an average of 9 months
  Identify FEV1 changes over time to characterize the pulmonary recovery trajectory of survivors of COVID-19.
FVC | Through study completion, an average of 9 months
  Identify FVC changes over time to characterize the pulmonary recovery trajectory of survivors of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Mylinh Duong, MD, Principal Investigator — McMaster University Hospital
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No